CLINICAL TRIAL: NCT05553717
Title: Clinical Study Evaluating the Gastroprotective Effect of Carvedilol in Patients With Ischemic Heart Disease on Aspirin Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sarah Mohamed Elkablawy, Clinical pharmacy master candidate, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: carvedilol as Gastroprotective
Record Dates: First submitted 2022-09-17; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: IHD; Gastro-Intestinal Disorder; Aspirin Induced Esophageal Ulcer
MeSH Terms: conditions — Digestive System Diseases | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): 33 patients who will receive aspirin 150mg + carvedilol 12.5mg twice daily plus other traditional therapy of ischemia for three months.
  Interventions: Drug: Carvedilol
- group 2 control (No Intervention): 33 patients who will receive aspirin 150mg + Captopril 12.5mg twice daily plus other traditional therapy of ischemia for three months.

INTERVENTIONS:
Drug: Carvedilol — Carvedilol 12.5mg\12hr
  Arms: group 1

SUMMARY:
The aim of this study is to investigate the possible efficacy of Carvedilol as gastroprotective agent against aspirin-induced upper gastro-intestinal complications in patients with ischemic heart disease (IHD).

DETAILED DESCRIPTION:
Gastric ulcer is a common gastrointestinal tract (GIT) disorder that affects about 4 million of the world's population annually, with incidence of complications in approximately 10%-20%. Gastric ulcer impacts negatively on the health-related quality of life of the affected individuals (1). It is characterized by GIT bleeding, perforation, and erosion of the mucosa wall due to imbalance between aggressive factors (acid, pepsin, and Helicobacter pylori) and defensive factors (mucin, prostaglandins (PG), bicarbonate, nitric oxide (NO), mucosal blood flow, and growth factors) (2). Most cases of peptic ulcer disease are associated with Helicobacter pylori infection or the use of nonsteroidal anti-inflammatory drugs (NSAIDs), or both (3). Aspirin or acetylsalicylic acid that has been used as analgesic, antipyretic and antiinflammatory agent against multiple types of inflammation and in the prevention of cardiovascular thrombotic diseases as myocardial infarction (4). Despite its therapeutic benefits, the use of aspirin is a major problem secondary to the associated risk for gastric ulcer (5). Low doses of aspirin were reported to be associated with gastric and duodenal ulcers (6-12). The pathogenesis of aspirin-induced gastric ulceration includes that, the aspirin inhibits the activities of the cyclooxygenase (COX) leading to decrease in prostaglandin (PG) with subsequent reduction in mucus and bicarbonate secretion, decreasing mucosal blood flow, impairment of platelet aggregation, alteration of microvascular structures leading to epithelia damage, increased leukocyte adherence and increased production of inflammatory mediators, reactive oxygen species (ROS) and decreased antioxidant enzymes (13). Enteric-coated aspirin has less gastrointestinal toxicity, but as compared to uncoated formulations, its plasma peak level after oral intake seems slower than traditional formulation (3 to 4 hours vs 15 to 20 minutes). In addition, enteric-coated aspirin is also associated with reduced bioavailability (14). Carvedilol is an antihypertensive agent that is commonly used in the treatment of arterial hypertension, heart failure, and angina pectoris based on its combined β- and α1- blocking activities. its therapeutic benefit also includes its antioxidant and antiperoxidative properties. It has been also shown that, carvedilol acts as a metal scavenger and can protect mitochondria against oxidative damage (15). Furthermore, carvedilol showed anti-oxidative and anti-inflammatory activities against renal, hepato, and cardiotoxicity. Additionally, it is hypothesized that carvedilol has protective effects against aspirin-induced gastric ulcer or gastrointestinal toxicity (16). Very few studies are present regarding the protective effects of Carvedilol on aspirin-induced gastric ulcer. A recent study revealed that, Carvedilol use was associated with an improvement in histopathological pictures of gastric ulcers in animals' model of cold stress ulcer (17).

The previously mentioned findings highlight the need for further studies to evaluate the role of carvedilol as gastroprotective in patient on aspirin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-60 years.
2. Both genders.
3. Patient with IHD including myocardial infarction, unstable angina and chronic stable angina on aspirin therapy.
4. Patients with hypertension.
5. Patients on low dose aspirin therapy for at least 3 months.

Exclusion Criteria:

1. Subjects with history of gastrointestinal disease, gastroduodenal surgery, H. pylori infection.
2. History or current diagnosis of major depressive disorder or other psychiatric disorders.
3. Patients already under histamine-2 receptor antagonist, proton pump inhibitor, misoprostol or gastrofate within 2 weeks of entering this study.
4. Patients who are allergic to aspirin and NSAIDs, who have an intolerance to aspirin and NSAIDs.
5. Subjects with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorders.
6. Pregnancy or lactation.
7. Patients with severe hepatic impairment (Child-Pugh class B and C) or total bilirubin level ≥ 1.2 mg/dl.
8. Patients with renal impairment (creatinine clearance less than 50mg/dl).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation the change in gastrointestinal symptoms. | 3 months
  improve gastrointestinal symptoms by assessment the change in SAGIS questionnaire
Quality of life of IHD patients | 3 months
  Improve quality of life according SAQ-7 questionair

SECONDARY OUTCOMES:
the changes in the measured biomarkers | 3 months
  Hydroxynonenal serum level , high level indicate gastric ulcer , using commercially available ELISA kit.
Change in PGE2 | 3 months
  High level of PGE2 indicate gastric mucosa integrity,using commercially available ELISA kit.
Change in Gastrin-17 serum . | 3 months
  Low level of gastrin-17 indicate high acid output ,using commercially available ELISA kit.
Malondialdehyde (MDA) serum level | 3months
  indicator of oxidative stress and can be measured in ulcerative and inflammatory conditions of the gastrointestinal tract, using commercially available method (colorimetric method).

REFERENCES:
- [Background] Kavitt RT, Lipowska AM, Anyane-Yeboa A, Gralnek IM. Diagnosis and Treatment of Peptic Ulcer Disease. Am J Med. 2019 Apr;132(4):447-456. doi: 10.1016/j.amjmed.2018.12.009. Epub 2019 Jan 3. PMID 30611829
- [Background] Patrono C, Baigent C. Role of aspirin in primary prevention of cardiovascular disease. Nat Rev Cardiol. 2019 Nov;16(11):675-686. doi: 10.1038/s41569-019-0225-y. Epub 2019 Jun 26. PMID 31243390
- [Background] Cadavid AP. Aspirin: The Mechanism of Action Revisited in the Context of Pregnancy Complications. Front Immunol. 2017 Mar 15;8:261. doi: 10.3389/fimmu.2017.00261. eCollection 2017. PMID 28360907
- [Background] Chitapanarux T, Lertprasertsuke N, Kongnak A. Teprenone for the prevention of low-dose aspirin-induced gastric mucosal injury in Helicobacter pylori-negative patients. Scand J Gastroenterol. 2019 Oct;54(10):1199-1204. doi: 10.1080/00365521.2019.1672781. Epub 2019 Oct 8. PMID 31591940
- [Background] Valkhoff VE, Sturkenboom MC, Hill C, Veldhuyzen van Zanten S, Kuipers EJ. Low-dose acetylsalicylic acid use and the risk of upper gastrointestinal bleeding: a meta-analysis of randomized clinical trials and observational studies. Can J Gastroenterol. 2013 Mar;27(3):159-67. doi: 10.1155/2013/596015. PMID 23516680
- [Background] Osman AS, Labib DA, Kamel MM. Carvedilol can attenuate histamine-induced paw edema and formaldehyde-induced arthritis in rats without risk of gastric irritation. Int Immunopharmacol. 2017 Sep;50:243-250. doi: 10.1016/j.intimp.2017.07.004. Epub 2017 Jul 12. PMID 28711030
- [Background] Ahmed I, Elkablawy MA, El-Agamy DS, Bazarbay AA, Ahmed N. Carvedilol safeguards against aspirin-induced gastric damage in rats. Hum Exp Toxicol. 2020 Sep;39(9):1257-1267. doi: 10.1177/0960327120918306. Epub 2020 Apr 15. PMID 32295429
- [Background] Koloski NA, Jones M, Hammer J, von Wulffen M, Shah A, Hoelz H, Kutyla M, Burger D, Martin N, Gurusamy SR, Talley NJ, Holtmann G. The Validity of a New Structured Assessment of Gastrointestinal Symptoms Scale (SAGIS) for Evaluating Symptoms in the Clinical Setting. Dig Dis Sci. 2017 Aug;62(8):1913-1922. doi: 10.1007/s10620-017-4599-6. Epub 2017 May 27. PMID 28551709
- [Background] Gierlaszynska K, Pudlo R, Jaworska I, Byrczek-Godula K, Gasior M. Tools for assessing quality of life in cardiology and cardiac surgery. Kardiochir Torakochirurgia Pol. 2016 Mar;13(1):78-82. doi: 10.5114/kitp.2016.58974. Epub 2016 Mar 30. PMID 27212988
- [Derived] Elkablawy SM, Shaban AE, Mostafa TM. Clinical study evaluating the gastroprotective effect of carvedilol in patients with ischemic heart disease on aspirin therapy. Inflammopharmacology. 2025 Nov;33(11):6831-6838. doi: 10.1007/s10787-025-01961-1. Epub 2025 Sep 30. PMID 41028410